CLINICAL TRIAL: NCT03231657
Title: Randomizated Open-label Control Trial to Evaluate if the Incorporation of sFlt1/PlGF Ratio in the Diagnosis and Classification of PE Improves Maternal and Perinatal Outcomes in Women With the Suspicion of the Disease (EuroPE Study)
Brief Title: Randomizated Open-label Control Trial to Evaluate if the Incorporation of sFlt1/PlGF Ratio in the Diagnosis and Classification of PE Improves Maternal and Perinatal Outcomes in Women With the Suspicion of the Disease
Acronym: EuroPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Carlos III Health Institute (Other Government); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-EUR-2017-20
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2022-08

CONDITIONS: Preeclampsia
Keywords: preeclampsia; intrauterine growth restriction; angiogenic factors
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incorporation of the sFlt1/P1GF ratio (Experimental): Incorporation of the ratio in the diagnosis and classification of pre-eclampsia:
  * sFlt1/PlGF ratio >38: pre-eclampsia risk
  * sFlt1/PlGF ratio >85: pre-eclampsia
  * ISSHP pre-eclampsia definition + ratio >210: severe PE
  * ISSHP pre-eclampsia definition + ratio sFlt1/PlGF ratio >600: consider deliver
  Interventions: Diagnostic Test: Placental biomarkers
- Routine clinical practice (No Intervention): Criteria for the definition of PE were those of the International Society for the Study of Hypertension in Pregnancy

INTERVENTIONS:
Diagnostic Test: Placental biomarkers — sFlt1 and P1GF levels and sFlt1/PlGF ratio
  Arms: Incorporation of the sFlt1/P1GF ratio

SUMMARY:
Preeclampsia is a leading cause of maternal and neonatal morbidity and mortality worldwide. The morbidity and mortality of this condition arises from two main causes: 1) the lack of specific and sensible methods for its diagnosis and prognosis, 2) and the fact that the course of the disease is often unpredictability at its presentation and speed of progression. The majority of deaths are undoubtedly avoidable and are due to a substandard care. Nowadays it's known that preeclampsia is a placental disorder that is characterized by an unbalance of angiogenic and antiangiogenic factors. It has been recently proven that the ratio of sFlt-1 to PlGF in women who presented with a clinical suspicion of preeclampsia is useful distinguishing between women in whom preeclampsia would develop and those in whom it would not. A low ratio also predicted the absence of fetal adverse outcomes in the same time frame. In addition this ratio demonstrated to be useful to discriminate among patients that would developed maternal or fetal adverse outcome. Correct identification and diagnosis of women at risk could potentially prevent all these adverse outcomes thus, clinical experience suggests that early detection and monitoring are beneficial.

EuroPE aims to provide evidence that the re-definition of pre-eclampsia as an entity caused by a placental unbalance of angiogenic and anti-angiogenic factors and its incorporation in the diagnosis and classification of the disease would improve maternal and neonatal health.

This will be an open, multicentre, international, randomised controlled trial with an intention-to -treat analysis. The study is pragmatic: it will be undertaken to reflect real clinical practice rather than the very tightly controlled circumstances of explanatory trials. The main objective of this study is to determine the effects of the use of the ratio as a diagnostic tool in the definition and classification of PE, as compared with its usual definition, in triage and delivery decisions and to see whether this new approach is able to improve maternal and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand informed consent.
* Unique pregnancies.
* > 24 weeks and <41 weeks
* Suspected preeclampsia:

  1. 140/90 or worsening of chronic hypertension
  2. Onset of proteinuria (Labstick + or proteinuria> 300mg / 24 hours) or worsening of it
  3. Preeclampsia prodromal clinic such as epigastric, headache, photopsia, tinnitus and increased edema in the face hands or legs or weight gain (> 1 kg per week in the third trimester)
  4. Analytical alterations: decrease in platelets <100,000. Increased transaminases.
  5. Ultrasound alterations: Small fetus for gestational age or restriction of interatrial growth, increased resistance of the uterine arteries.
* Pre-eclampsia (ACOG Practice Bulletin 2013)

Exclusion Criteria:

* Multiple pregnancies
* <24 weeks of gestation
* Fetal chromosomal or congenital abnormalities
* Conditions that require immediate delivery (eclampsia, pulmonary edema, uncontrolled hypertension, severe visual disturbances, severe headache, fetal demise, non-reassuring fetal status….)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2536 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Adverse outcomes | Up to 24 weeks
  Composite score for adverse outcomes defined as the presence of any of the following: premature placental abruption, cessation of abnormal CTG, fetal death, need for 2 or more antihypertensive drugs, eclampsia, disseminated intravascular coagulation, maternal mortality, postpartum haemorrhage (need for more than 2 concentrated hematies), acute pulmonary edema, cerebral vascular hemorrhage, pulmonary embolism, sepsis, ICU admission, need for second surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990
- [Background] Verlohren S, Herraiz I, Lapaire O, Schlembach D, Zeisler H, Calda P, Sabria J, Markfeld-Erol F, Galindo A, Schoofs K, Denk B, Stepan H. New gestational phase-specific cutoff values for the use of the soluble fms-like tyrosine kinase-1/placental growth factor ratio as a diagnostic test for preeclampsia. Hypertension. 2014 Feb;63(2):346-52. doi: 10.1161/HYPERTENSIONAHA.113.01787. Epub 2013 Oct 28. PMID 24166751
- [Background] von Dadelszen P, Payne B, Li J, Ansermino JM, Broughton Pipkin F, Cote AM, Douglas MJ, Gruslin A, Hutcheon JA, Joseph KS, Kyle PM, Lee T, Loughna P, Menzies JM, Merialdi M, Millman AL, Moore MP, Moutquin JM, Ouellet AB, Smith GN, Walker JJ, Walley KR, Walters BN, Widmer M, Lee SK, Russell JA, Magee LA; PIERS Study Group. Prediction of adverse maternal outcomes in pre-eclampsia: development and validation of the fullPIERS model. Lancet. 2011 Jan 15;377(9761):219-27. doi: 10.1016/S0140-6736(10)61351-7. Epub 2010 Dec 23. PMID 21185591
- [Background] National Institute for Health and Care Excellence guideline DG 23 (2016): PlGF based testing to help diagnose suspected pre-eclampsia (Triage PlGF test, Elecsys immunoassay sFlt-1/PlGF ratio, DELFIA Xpress PlGF 1-2-3 test, and BRHAMS sFlt-1 Kryptor/BRAHMS PlGF plus Kryptor PE ratio). Available at: https://www.nice.org.uk/guidance/dg23/chapter/1-recommendations [Accessed January 2017].
- [Background] Stepan H, Herraiz I, Schlembach D, Verlohren S, Brennecke S, Chantraine F, Klein E, Lapaire O, Llurba E, Ramoni A, Vatish M, Wertaschnigg D, Galindo A. Implementation of the sFlt-1/PlGF ratio for prediction and diagnosis of pre-eclampsia in singleton pregnancy: implications for clinical practice. Ultrasound Obstet Gynecol. 2015 Mar;45(3):241-6. doi: 10.1002/uog.14799. No abstract available. PMID 25736847